CLINICAL TRIAL: NCT01226615
Title: Randomized, Double-blind, Placebo-controlled Study to Asses the Effect of Chondroitin Sulphate in Patients With Knee Osteoarthritis by Functional Magnetic Resonance Imaging
Brief Title: Assessment of the Effects of Chondroitin Sulphate in Patients With Knee Osteoarthritis With Functional Magnetic Resonance Imaging (fMRI)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bioiberica (Industry)
Responsible Party: Dr. Josep Vergés, Scientific Medical Director, Bioibérica S.A.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CS/IV-RMF-01
Record Dates: First submitted 2010-10-08; First posted 2010-10-22 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Knee Osteoarthritis
Keywords: Chondroitin sulphate; Knee osteoarthritis; Functional Magnetic Resonance Imaging
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Chondroitin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Chondroitin sulphate
  Interventions: Drug: Chondroitin sulphate (Condrosan®)
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chondroitin sulphate (Condrosan®) — 800mg (two capsules of 400mg each) taken once a day for four months
  Arms: 1
Drug: Placebo — Two placebo capsules taken once a day for four months.
  Arms: 2

SUMMARY:
The main purposes of this study are:

* to determine the effects of chondroitin sulphate on brain response to pain assessed through fMRI in patients with knee osteoarthritis.
* to investigate the relationship between treatment response detected by fMRI and the results of the different parameters of clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

* Primary knee OA according to ACR criteria
* OA of radiological stages 2 to 3 according to Kellgren-Lawrence
* Estable knee pain during the last months before to start the clinical trial
* Patients with pain as the VAS≥50mm at baseline

Exclusion Criteria:

* Patients with skin conditions that could interfere in the clinical trial evaluation
* Pregnant or breastfeeding woman
* Patients with a history of alcoholism or other drug abuse
* Patients with an uncontrolled active psychiatric disorder
* Patients with other inflammatory or systemic conditions affecting other joints
* Patients who suffer more intense pain in the joint in another location
* Patients unable to differentiate between symptoms caused by the knee in front of the joint study opposite
* OA of radiological stages 1 or 4 according to Kellgren-Lawrence
* Other bone and articular diseases such as chondrocalcinosis, Paget's disease, rheumatoid arthritis, aseptic osteonecrosis, gout, septic arthritis, ochronosis, acromegaly, hemochromatosis, Wilson's disease, osteochondromatosis
* Patients with contraindications to perform an MRI such as: certain tattoos, pacemakers, intracranial clips incompatible with MRI, in the heart valves, hearing aids and other types of implants are incompatible with MRI
* Known allergy to chondroitin sulphate
* Washout period for OA treatments before beginning the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Brain response to pain caused on arthritic knee selected by fMRI | 4 months
  Functional magnetic resonance imaging (fMRI) is particularly suited to investigating the effects of pharmacological agents on pain processing within the human central nervous system.
  The measures are based on the haemodynamic resonse to a neuronal event and constitute indirect measures of excitatory and inhibitory neuronal activity. The neuronal activation is associated with an increase of the oxygen extraction fraction from the capillaries and with an increase in regional cerebral blood flow. The measure which derived from blood oxygenation is called the BOLD effect.

SECONDARY OUTCOMES:
Assessment of the reduction of pain by Huskisson VAS | 4 months
Determination of pain and functional capacity using the Lequesne Algofunctional Index | 4 months
Use of rescue medication | 4 months
Assessment of the quality of life of patients by SF-36 Health Questionaire | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Monfort, MD, Principal Investigator — Hospital del Mar; Jesús Pujol, MD, Principal Investigator — Hospital del Mar
Locations (1):
- Hospital del Mar, Barcelona, Barcelona, Spain